CLINICAL TRIAL: NCT02969304
Title: Claims Database Study of Utilization Patterns of Dimethyl Fumarate in Germany
Brief Title: Study of Utilization Patterns of Dimethyl Fumarate in Germany
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 109MS409
Record Dates: First submitted 2016-10-21; First posted 2016-11-21 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Multiple Sclerosis
Keywords: Tecfidera; Off-label; Utilization
MeSH Terms: conditions — Multiple Sclerosis; Patient Acceptance of Health Care | interventions — Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Off-Label: Any DMF prescription for MS patients <18 years of age, or for patients diagnosed with non-MS indications, such as psoriasis.
  Interventions: Drug: dimethyl fumarate
- On-Label: Prescriptions for patients who are ≥18 years of age and diagnosed with MS
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — Off-Label Use: All participants <18 years of age and participants without an MS diagnosis who are prescribed dimethyl fumarate
  On-Label Use: All participants >18 years of age with an MS diagnosis who are prescribed dimethyl fumarate
  Other Names: Tecfidera, DMF, BG00012

SUMMARY:
The primary objective of this study is to estimate the proportion of DMF use that is prescribed "on-label" versus "off-label". The secondary objectives are: To describe the demographic characteristics and medical history of DMF users; To describe prescription drug history and concomitant medication use of DMF users; To describe the duration of therapy in participants newly initiating DMF treatment; To describe the medical specialties of DMF prescribers.

DETAILED DESCRIPTION:
Dimethyl fumarate will not be provided to participants as a part of this study.

ELIGIBILITY:
Key Inclusion Criteria:

* New users of dimethyl fumarate will be included in the analysis

Key Exclusion Criteria:

* Patients for which data is not available for the 6 months period prior to the index date (baseline observational period)

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective analysis of a research database, which contains German sick fund claims, to assess the usage of dimethyl fumarate in Germany. The research database is comprised of German sick fund data, which is compiled by Gesundheitsforen Leipzig (GFL). This GFL database currently contains sick fund claims data for approximately 4 million patients, which accounts for approximately 5-6% of the total sick fund population in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 930 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Proportion of dimethyl fumarate use that is prescribed "on-label" versus "off-label" in Germany | Up to 18 months after market introduction of dimethyl fumarate in Germany

SECONDARY OUTCOMES:
Demographic characteristics of dimethyl fumarate users | Up to 18 months after market introduction of dimethyl fumarate in Germany
Prescription drug history of dimethyl fumarate users | Up to 18 months after market introduction of dimethyl fumarate in Germany
Duration of therapy in participants newly initiating dimethyl fumarate treatment | Up to 18 months after market introduction of dimethyl fumarate in Germany
Number of medical specialists prescribing dimethyl fumarate as identified according to specialty-specific billing codes at outpatient visits. | Up to 18 months after market introduction of dimethyl fumarate in Germany
Medical history of dimethyl fumarate users | Up to 18 months after market introduction of dimethyl fumarate in Germany
Concomitant medication use of dimethyl fumarate users | Up to 18 months after market introduction of dimethyl fumarate in Germany

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Leipzig, Saxony, Germany